CLINICAL TRIAL: NCT03497325
Title: the Efficacy of Intramuscular Autologous Platelet-rich Plasma Injection on Uterine Wound Healing After Primary Cesarean Section
Brief Title: Effect of Autologous Platelet-rich Plasma in Uterine Wound Healing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASUM hospital
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP (Experimental): 55 participant unergoing prelabor primary CS will receive intramyometrial injection of PRP after closure of uterine incision
  Interventions: Drug: autologus platelet rich plasma
- placebo (Placebo Comparator): 55 participant unergoing prelabor primary CS will receive intramyometrial injection of normal saline after closure of uterine incision
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: autologus platelet rich plasma — 55 participant unergoing prelabor primary CS will receive intramyometrial injection of PRP after closure of uterine incision
  Arms: PRP
Drug: placebo — 55 participant unergoing prelabor primary CS will receive intramyometrial injection of normal saline after closure of uterine incision
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate the efficacy of intramuscular autologus platelet rich plasma on uterine wound healing after primary cesarean section

DETAILED DESCRIPTION:
110 pregnant female undergoing primary prelabor CS will be randomized to two groups group A)autologus PRP will be prepared from participant venous blood collected from the participants' arm into a syringe primed with ACD-A. then it will be injected into uterus after closing uterine incision . Injection sites will be selected near the incision at evenly 20 different sites

group B)normal saline 0.9 will be injected into uterus after closing uterine incision . Injection sites will be selected near the incision at evenly 20 different sites.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy (gestational age between 37-41 weeks).
* Women undergoing cesarean section for the first time.
* Normal vaginal ultrasound examination and exclusion of any pelvic abnormality.
* Uncomplicated cesarean section.
* Lower uterine segment cesarean sections while the women not in labor

Exclusion Criteria:

* Women with complications during or after cesarean section as intrapartum or postpartum hemorrhage, puerperal sepsis, septic wound
* Women with medical diseases that can affect the healing as diabetes mellitus, anemia, chronic renal disease or hepatic disease or coagulopathy or receiving medications affect wound healing as corticosteroids or anticoagulant.
* Women who will use intrauterine device as a contraceptive method Women with uterine abnormality as cervical stenosis or fibroid uterus multiple gestation, placenta abruption, placenta previa, antepartum hemorrhage prolonged ROM, chorioamnionitis,meconium stained liquor

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Presence of cesarean scar defect(niche) | 12 weeks after CS
  any defect in the anterior myometrium related to scar site

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university maternity hospital, Cairo, Egypt